CLINICAL TRIAL: NCT02087865
Title: Effects of Donepezil HCL on Task-Activated fMRI Brain Activation in Healthy Older Adults at Genetic Risk for Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Stephen Rao, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 14-227
Record Dates: First submitted 2014-03-07; First posted 2014-03-14 (Estimated); Results first posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Genetic Risk for Alzheimer's Disease
MeSH Terms: interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Donepezil HCL (Active Comparator): Participants will receive 5mg of donepezil HCL for 4 weeks and then 10mg of donepezil HCL for 20 weeks.
  Interventions: Drug: donepezil HCL
- Placebo (Placebo Comparator): Participants will receive placebo for 24 weeks.
  Interventions: Drug: Placebo
- Control Group (No Intervention): Participants without a family history of AD will undergo the study evaluations but will not receive any study drug

INTERVENTIONS:
Drug: donepezil HCL
  Arms: Donepezil HCL
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study examines the sensitivity of functional MRI to detect brain changes caused by donepezil HCL (a cholinesterase inhibitor) in healthy older adults at genetic risk for Alzheimer's Disease.

DETAILED DESCRIPTION:
This 24-week study will examine the sensitivity of functional MRI to detect brain changes caused by donepezil HCL (a cholinesterase inhibitor) in healthy older adults at genetic risk for Alzheimer's Disease. Participants with a family history of Alzheimer's Disease will be eligible for this study. Participants without a family history of AD will also be enrolled to serve as a control group.

ELIGIBILITY:
Inclusion Criteria:

* Normal general cognitive function
* High Risk Group Only: Family history (1st degree relative) of AD
* Low Risk Group Only: No family history (1st or 2nd degree relative) of AD
* Visual and auditory acuity adequate for neuropsychological testing

Exclusion Criteria:

* Current or past history of
* neurological illnesses/conditions
* head trauma with significant loss of consciousness
* medical illnesses/conditions that may affect brain function
* severe psychiatric disorder
* substance abuse
* unstable or severe cardiovascular disease or asthmatic condition
* history of stroke or transient ischemic attack

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Rao, Ph.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Center for Brain Health, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Donepezil HCL: Participants will receive 5mg of donepezil HCL for 4 weeks and then 10mg of donepezil HCL for 20 weeks.
  donepezil HCL
- Placebo: Participants will receive placebo for 24 weeks.
  Placebo
Period: Overall Study
Arm/Group | Donepezil HCL | Placebo | Control Group
Started | 28 | 29 | 32
Completed | 22 | 26 | 29
Not Completed | 6 | 3 | 3
Not completed — Withdrawal by Subject | 6 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Drug Non-compliance | 0 | 2 | 0
Not completed — Not analyzed due to anatomical abnormalities | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The number reflects the participants who completed the study in the respective study groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil HCL | Placebo | Control Group | Total
Number analyzed (Participants) | 22 | 26 | 29 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 9 | 11 | 26
  >=65 years | 16 | 17 | 18 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (4.1) | 66.1 (3.8) | 67.7 (4.7) | 66.8 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 18 | 48
  Male | 6 | 12 | 11 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 26 | 28 | 76
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 6
  White | 21 | 21 | 27 | 69
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 26 | 29 | 77

OUTCOME MEASURES:

1. Primary Outcome: Change in BOLD Response From Baseline to 24 Weeks During Functional Magnetic Resonance Imaging - Left Posterior Cingulate BOLD Signal at 24 Weeks, Adjusting for Baseline Left Posterior Cingulate BOLD
Description: Changes from baseline to 24 weeks follow-up fMRI - Left posterior cingulate BOLD signal at 24 weeks, adjusting for baseline left posterior cingulate BOLD signal.
Time Frame: Baseline and 24 Weeks
Population: Please note that the fMRI result of one subject was collected but could not be processed due to data quality issues. Hence, only 21 subjects in Donepezil HCL arm were analyzed.
Measure: Mean (Standard Deviation); unit: 100 * % Signal Change
Arm/Group | Donepezil HCL | Placebo | Control Group
Number analyzed (Participants) | 21 | 26 | 29
100 * % Signal Change | 44.68 (33.86) | 50.61 (23.46) | 45.57 (25.24)
Statistical Analysis 1: Comparison: Donepezil HCL vs Placebo; We are reporting the difference in mean between the Donepezil HCL and Placebo groups; Test type: Superiority; p = 0.273, ANCOVA; Mean Difference (Final Values) = -8.25, 95% CI 2-sided [-23.12 to 6.63], Standard Error of Mean 7.59

2. Primary Outcome: Left Hippocampus BOLD Signal at 24 Weeks, Adjusted for Baseline Left Hippocampus BOLD Signal
Description: Left hippocampus BOLD signal at 24 weeks, adjusting for baseline left hippocampus BOLD signal.
Time Frame: Baseline and 24 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 100 * % Signal Change
Arm/Group | Donepezil HCL | Placebo | Control Group
Number analyzed (Participants) | 21 | 26 | 29
100 * % Signal Change | 19.91 (8.69) | 32.31 (16.62) | 19.38 (14.02)
Statistical Analysis 1: Comparison: Donepezil HCL vs Placebo; We are reporting the difference in mean between the Donepezil HCL and Placebo groups; Test type: Superiority; p = 0.001, ANCOVA; Mean Difference (Final Values) = -13.41, 95% CI 2-sided [-21.09 to -5.73], Standard Error of Mean 3.92

3. Primary Outcome: Right Hippocampus BOLD Signal at 24 Weeks, Adjusted for Baseline Left Hippocampus BOLD Signal
Description: Right hippocampus BOLD signal at 24 weeks, adjusting for baseline left hippocampus BOLD signal.
Time Frame: Baseline and 24 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 100 * % Signal Change
Arm/Group | Donepezil HCL | Placebo | Control Group
Number analyzed (Participants) | 21 | 26 | 29
100 * % Signal Change | 24.9 (18.72) | 32.78 (20.57) | 26.73 (18.09)
Statistical Analysis 1: Comparison: Donepezil HCL vs Placebo; We are reporting the difference in mean between the Donepezil HCL and Placebo groups; Test type: Superiority; p = 0.115, ANCOVA; Median Difference (Final Values) = -8.60, 95% CI 2-sided [-19.33 to 2.14], Standard Error of Mean 5.48

4. Secondary Outcome: Neuropsychological Testing Scores - Rey Auditory Verbal Learning Test (RAVLT) Sum of Trials (1-5) at 24 Weeks, Adjusted for Baseline RAVLT Score
Description: Rey Auditory Verbal Learning Test (RAVLT) (Sum of Trials 1-5) , adjusting for baseline RAVLT (Sum of Trials 1-5) score. The RAVLT total score has a minimum of 0 and a maximum of 75 correct items (15 per trial x 5 trials). A higher score means better outcomes.
Time Frame: Baseline and 24 Weeks
Measure: Mean (Standard Deviation); unit: Total number of correct items
Arm/Group | Donepezil HCL | Placebo | Control Group
Number analyzed (Participants) | 22 | 26 | 29
Total number of correct items | 52.86 (7.76) | 53.58 (9.71) | 51.41 (7.40)
Statistical Analysis 1: Comparison: Donepezil HCL vs Placebo; We are reporting the difference in mean between the Donepezil HCL and Placebo groups; Test type: Superiority; p = 0.941, ANCOVA; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-3.94 to 4.25], Standard Error of Mean 2.09

5. Secondary Outcome: Left Hippocampus Volume (MRI) at 24 Weeks, Adjusted for Baseline Left Hippocampus Volume
Description: Left hippocampus volume (MRI) at 24 weeks, adjusting for baseline left hippocampus volume
Time Frame: Baseline and 24 Weeks
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Donepezil HCL | Placebo | Control Group
Number analyzed (Participants) | 22 | 26 | 29
mm^3 | 3309.51 (300.08) | 3289.36 (260.1) | 3296.68 (312.89)
Statistical Analysis 1: Comparison: Donepezil HCL vs Placebo; We are reporting the difference in mean between the Donepezil HCL and Placebo groups; Test type: Superiority; p = 0.003, ANCOVA; Mean Difference (Final Values) = 46.33, 95% CI 2-sided [16.14 to 76.53], Standard Error of Mean 15.40

6. Secondary Outcome: Right Hippocampus Volume (MRI) at 24 Weeks, Adjusted for Baseline Right Hippocampus Volume
Description: Right hippocampus volume (MRI) at 24 weeks, adjusting for baseline right hippocampus volume
Time Frame: Baseline and 24 Weeks
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Donepezil HCL | Placebo | Control Group
Number analyzed (Participants) | 22 | 26 | 29
mm^3 | 1810.88 (231.08) | 1756.92 (183.39) | 3363.62 (214.59)
Statistical Analysis 1: Comparison: Donepezil HCL vs Placebo; We are reporting the difference in mean between the Donepezil HCL and Placebo groups; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 61.36, 95% CI 2-sided [35.25 to 87.46], Standard Error of Mean 13.32

7. Secondary Outcome: Brief Visuospatial Memory Test (BVMT) Learning Scores at 24 Weeks, Adjusted for Baseline BVMT Learning Scores
Description: Brief Visuospatial Memory Test (BVMT) learning scores at 24 weeks, adjusted for baseline BVMT learning scores. The BVMT-R total scare has a minimum of 0 and a maximum of 36 correct items (12 per trial x 3 trials). A higher score means better outcomes.
Time Frame: Baseline and 24 Weeks
Measure: Mean (Standard Deviation); unit: Total number of correct items
Arm/Group | Donepezil HCL | Placebo | Control Group
Number analyzed (Participants) | 22 | 26 | 29
Total number of correct items | 21.41 (6.17) | 23.58 (5.84) | 23.28 (5.07)
Statistical Analysis 1: Comparison: Donepezil HCL vs Placebo; We are reporting the difference in mean between the Donepezil HCL and Placebo groups; Test type: Superiority; p = 0.005, ANCOVA; Mean Difference (Final Values) = -3.35, 95% CI 2-sided [-5.65 to -1.04], Standard Error of Mean 1.18

8. Secondary Outcome: Processing Speed Test (PST) at 24 Weeks, Adjusted for Baseline PST Scores
Description: Processing speed test (PST) at 24 weeks, adjusting for baseline PST scores. The PST has a minimum of 0 and no upper limit/maximum since it is the number of correct items in 2 minutes. A higher score means better outcome.
Time Frame: Baseline and 24 Weeks
Population: Please note only those participants who had complete PST data were included in the analysis, which are 12 participants in Donepezil HCL group, 15 participants in Placebo group, and 22 participants in Control group.
Measure: Mean (Standard Deviation); unit: Total number of correct items
Arm/Group | Donepezil HCL | Placebo | Control Group
Number analyzed (Participants) | 12 | 15 | 22
Total number of correct items | 44.17 (7.96) | 49.8 (4.69) | 47.73 (4.87)
Statistical Analysis 1: Comparison: Donepezil HCL vs Placebo; We are reporting the difference in mean between the Donepezil HCL and Placebo groups; Test type: Superiority; p = 0.011, ANCOVA; Mean Difference (Final Values) = -4.30, 95% CI 2-sided [-7.58 to -1.02], Standard Error of Mean 1.67

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Donepezil HCL | Placebo | Control Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29 | 0/32
Other Adverse Events (participants affected / at risk) | 20/28 | 13/29 | 0/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil HCL (N=28) | Placebo (N=29) | Control Group (N=32)
Nausea (General disorders) | 4 (4) | 0 (0) | 0 (0)
Dizziness (General disorders) | 4 (4) | 1 (1) | 0 (0)
Muscle cramping (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (2) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 0 (0)
Vivid dreams/Nightmares/Increased Dreams (General disorders) | 10 (11) | 1 (1) | 0 (0)
Loose stool/Diarrhea/Increased Bowel Movement (Gastrointestinal disorders) | 7 (7) | 3 (3) | 0 (0)
Rumbling stomach (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Disturbed sleep (General disorders) | 7 (8) | 0 (0) | 0 (0)
Persistent ringing in ears (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Recurrence of skin cancer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Decrease in appetite (General disorders) | 1 (1) | 2 (2) | 0 (0)
Fall (General disorders) | 2 (2) | 0 (0) | 0 (0)
Anxiety (General disorders) | 2 (2) | 0 (0) | 0 (0)
Change in vision/Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Mood changes/Mood swing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Frequent urge to urinate (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Increased talkativeness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lower than normal heart rate (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Altered liver function tests (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Change in consistency of saliva (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Headache/Pain in head or neck area (General disorders) | 1 (1) | 3 (3) | 0 (0)
Excessive thirts (General disorders) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Change in sexual intercourse or libido (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Hand surgery under general anesthesia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Scrotal blisters (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Paresthesia in legs (numbness, tingling sensation) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Change in facial skin color (Darker skin in cheek area) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Increase in size of colloid cyst with early signs of hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Change in sweat/body smell (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eyebrows falling out (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Kidney stones (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT02087865/Prot_SAP_000.pdf